CLINICAL TRIAL: NCT05596552
Title: Comparison of Intrathecal Dexmedetomidine Versus Fentanyl as Adjuvants to Bupivacaine on Post-operative Urinary Retention in Knee Joint Arthroscopic Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada M.Samir, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MS532/2021
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Post-Op Complication
MeSH Terms: conditions — Postoperative Complications | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine-Dexmedetomidine group (Active Comparator)
  Interventions: Drug: hyperbaric bupivacaine and dexmedetomidine
- Bupivacaine-Fentanyl group (Active Comparator)
  Interventions: Drug: Bupivacaine-Fentanyl group

INTERVENTIONS:
Drug: hyperbaric bupivacaine and dexmedetomidine — In a 3 ml syringe, 5 µg dexmedetomidine was added to the 2 ml of 10 mg hyperbaric bupivacaine, to have a total volume of 2.5 ml for intrathecal spinal injection over 3 minute without barbotage
  Arms: Bupivacaine-Dexmedetomidine group
Drug: Bupivacaine-Fentanyl group — In a 3 ml syringe, 25 μg fentanyl was added to the 2 ml of 10 mg hyperbaric bupivacaine, to have a total volume of 2.5 ml for intrathecal spinal injection over 3 minute without barbotage
  Arms: Bupivacaine-Fentanyl group

SUMMARY:
The aim of this study was to assess the effect of intrathecally injected 5 µg dexmedetomidine or 25 µg fentanyl as adjuvants to bupivacaine in low dose spinal anesthesia for unilateral arthroscopic knee surgeries, on post-operative urinary retention (POUR), time needed to reach sensory block at the tenth thoracic dermatome (T10), the maximum sensory level achieved, the onset of motor block, the intra-operative fluids given, the duration of sensory and motor blocks, time to micturition or insertion of an intermittent urinary catheter and the number of patients who needed an indwelling (Foley's) catheter. Seventy patients, ASA physical status I or II, from 21 to 50 years old, scheduled to undergo unilateral arthroscopic knee surgeries under spinal anesthesia, were randomly divided into two equal groups; the Bupivacaine- Dexmedetomidine group (BD) patients and the Bupivacaine-Fentanyl group (BF) patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II
* aged 21-50 years
* scheduled to undergo unilateral arthroscopic knee surgeries under spinal anesthesia

Exclusion Criteria:

* Patients' refusal
* contraindications to spinal anesthesia
* patients with coagulopathy
* infection at the lumbar region
* pre-existing neurological deficits in the lower limbs
* known allergy to any of the study drugs
* urinary incontinence
* cysto-ureteric reflux
* patients with congestive heart failure
* patients with dysrhythmia
* patients with heart block
* diabetic patients
* patients on α2-adrenergic receptors antagonists
* calcium channel blockers

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Post-operative urinary retention | 3 hours
  Ultrasound assessment of the urinary bladder volume was done at the 3rd post-operative hour, a bladder volume of >700 ml with no ability to void confirmed the presence of urinary retention

SECONDARY OUTCOMES:
Time to reach sensory block at T10 | 30 minutes
  The time from completion of intrathecal injection of the study drug till loss of sensation to pin prick at T10 on the operative side, assessed every 2 minutes.
Maximum sensory level achieved | 30 minutes
  Sensory level assessment by loss of sensation to pinprick every 2 minutes, until the highest level had stabilized for four consecutive tests
The onset of motor block | 30 minutes
  The time from completion of intrathecal injection of the study drug till having a modified Bromage score = 1 or more
Intra-operative fluids given | 3 hours
  The volume of IV Ringer's solution given to each patient according to the fluid chart
Duration of sensory block | 6 hours
  he time from completion of intrathecal injection of the study drug till regression to the third sacral dermatome (S3) level
Duration of motor block | 6 hours
  The time from completion of intrathecal injection of the study drug till complete recovery of the motor function (MBS = 0), by asking the patient to flex the hip, knee and ankle joints, in the PACU, then every 15 minutes in the ward
Time to micturition or insertion of an intermittent urinary catheter | 6 hours
  The time from completion of intrathecal injection of the study drug till voiding or insertion of an in-out catheter
Number of patients who needed an indwelling (Foley's) catheter | 6 hours
  After 6 post-operative hours, if the patient wasn't able to void an indwelling (Foley's) catheter was then placed

CONTACTS AND LOCATIONS:
Overall Officials: Ghada M Samir, MD, Principal Investigator — Faculty of Medicine, Ain- Shams University
Locations (1):
- Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided